CLINICAL TRIAL: NCT02602639
Title: Development of a Spinal Cord Injury-specific Exercise-based Capacity
Brief Title: Functional Electrical Stimulation With Rowing as Exercise After Spinal Cord Injury
Acronym: FES
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: University of Manitoba (Other)
Responsible Party: Principal Investigator, Kristine Cowley, Assistant Professor, University of Manitoba
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: H2014:174
Record Dates: First submitted 2015-11-05; First posted 2015-11-11 (Estimated); Last update posted 2020-06-26 (Actual); Status verified 2020-06

CONDITIONS: Spinal Cord Injury; Paraplegia; Tetraplegia
MeSH Terms: conditions — Spinal Cord Injuries; Paraplegia; Quadriplegia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Functional electrical stimulation rowing (Experimental): Using an Odstock 4 channel neuromuscular stimulator with Concept 2 Rower
  Interventions: Device: Functional electrical stimulation rowing (Odstock 4 channel neuromuscular stimulator with Concept 2 Rower)

INTERVENTIONS:
Device: Functional electrical stimulation rowing (Odstock 4 channel neuromuscular stimulator with Concept 2 Rower) — Participants will strengthen their quadriceps and hamstrings using electrical stimulation for up to 12 weeks (using an Odstock 4 channel neuromuscular stimulator). Then participants will use a seated rower (Concept 2 Rower, fitted with a backrest that allows those with spinal cord injury to engage in rowing) in conjunction with the electrical stimulation for 12-24 weeks.

SUMMARY:
Currently, those with spinal cord injury (SCI) demonstrate increased prevalence of obesity (75%) cardiovascular disease (30 - 50%), type II diabetes (21%) and osteoporosis in the legs (100%) when compared to the general population. It is important to identify the modes and intensities of exercise most likely to generate a reduction in these inactivity-related diseases in this population.

Therefore, the main purpose of this pilot research project is to implement and test a form of a spinal cord injury-specific exercise, known as FES rowing (FES: functional electrical stimulation).

ELIGIBILITY:
Inclusion Criteria:

* Have a spinal cord injury, C5-T12 (level), AIS A-D (severity)
* Be aged 18-75 for duration of study
* Medically stable and healthy enough to complete exercise requirements
* Willing and able to complete the at-home training requirements as prescribed
* Willing and able to complete the exercise sessions as prescribed
* Willing and able to complete the VO2 testing throughout the study
* Willing and able to complete the DEXA (Dual-energy X-ray absorptiometry) scans during the study
* Able to understand and follow written or verbal instructions from study staff

Exclusion Criteria:

* Current pressure ulcer(s) at sites of electrical stimulation
* Previous spontaneous or low-impact leg fracture
* Previous diagnosis of cardiovascular disease (ie enlarged heart, heart murmur)
* Unsatisfactory results of EKG (electrocardiogram) screening test
* Known thyroid dysfunction
* Kidney disease
* Cancer
* Blood pressure > 140/90 mmHg
* Currently taking blood pressure medication
* History of epilepsy
* Current hand, arm or shoulder injury
* Current deep vein thrombosis
* Implanted electronic cardiac device (pace maker, defibrillator, etc)
* Ventilator-dependent
* Unable to follow written and verbal instructions

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Estimated)
Dates: Start 2015-10 (Actual); Primary Completion 2021-12 (Estimated); Study Completion 2022-09 (Estimated)

PRIMARY OUTCOMES:
Peak VO2 (volume oxygen) output during exercise | 24 weeks compared to baseline
  Peak VO2 testing will be performed before beginning rower training and again at the end of the 24 weeks of training. Testing will be performed with an arm ergometer, rowing without electrical stimulation, and rowing with electrical stimulation. This will assess energy use, time to fatigue, and perceived exertion.

SECONDARY OUTCOMES:
Body composition | 24 weeks compared to baseline
  Participants will have their body composition (specifically leg percent fat and muscle, and bone mineral density) measured before beginning training and at the end of the 24 weeks of training.
Leg EMG (electromyogram) while rowing | Throughout study (up to 36 weeks)
  Participants will perform the rowing exercise while having EMG of multiple leg muscles.

CONTACTS AND LOCATIONS:
Overall Officials: Kristine Cowley, PhD, Principal Investigator — University of Manitoba
Locations (1):
- University of Manitoba, Winnipeg, Manitoba, Canada